CLINICAL TRIAL: NCT01164449
Title: Monocentric, Open Study to Investigate the Usability of Blood Glucose Control With the Space TGC System (With Incorporated Software-algorithm eMPC) Over a Glucose Control Range of 4.4 to 8.3 mmol/L in Medical ICU Patients
Brief Title: Usability of Blood Glucose Control With the Space TGC System in Medical ICU Patients
Acronym: DELIOS 4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Study Manager, B. Braun Melsungen AG
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HC-G-H-0910
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Critical Illness
Keywords: algorithm; tight glycemic control; glucose control; intensive care; insulin; ICU
MeSH Terms: conditions — Critical Illness; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Space TGC system with incorporated eMPC advised insulin titration to establish glycaemic control
  Interventions: Device: Space TGC

INTERVENTIONS:
Device: Space TGC — Space TGC with incorporated eMPC algorithm to establish glycaemic control with a blood glucose target range of 80-150 mg/dL (4.4-8.3 mM)

SUMMARY:
Hyperglycemia is common in critically ill patients and associated with an adverse outcome. Thus, glycaemic control is an important issue in critical care. Despite extensive efforts of the intensive care unit staff difficulties were experienced in achieving efficient and safe glucose control. A fully automated algorithm may help to overcome some of these limitations by excluding intuitive interventions and integrating relevant clinical data in the decision-making process. Space GlucoseControl (TGC system) is a decision support system which helps to achieve safe and reliable blood glucose control in the desired ranges. Information on parenteral and enteral nutrition is automatically integrated into the calculations. The primary objective of the current study is to investigate the performance and usability of the Space TGC system for glucose control in medical ICU patients.

ELIGIBILITY:
Inclusion:

* Age: > 18 years of age
* Stay in the ICU expected to be > 72 h
* Blood glucose > 6.1 mmol/L or patient on insulin treatment

Exclusion:

* Patients with hyperglycaemic crisis/ketoacidosis due to insulin deficiency.
* Known or suspected allergy to insulin
* Any disease or condition which the investigator or treating physician feels would interfere with the trial or the safety of the patient (i.e., liver failure, other fatal organ failures)
* Moribund patients likely to die within 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
(arterial) blood glucose values -> percentage of time within predefined glucose target range 80-150 mg/dL (4.4-8.3 mM) | all blood glucose measurements from start of treatment until last glucose measurement under treatment (i.e. stop of intravenous insulin treatment) up to a maximum of 14d

SECONDARY OUTCOMES:
Hypoglycaemia ≤ 40 md/dL (2.2mM) | all blood glucose measurements from start of treatment until last glucose measurement under treatment (i.e. stop of intravenous insulin treatment) up to a maximum of 14d
Usability parameters like convenience of alarming function; workload; blood sampling frequency | all blood glucose measurements from start of treatment until last glucose measurement under treatment (i.e. stop of intravenous insulin treatment) up to a maximum of 14d
Concomitant medication including insulin infusion rate, parenteral/enteral nutrition | all blood glucose measurements from start of treatment until last glucose measurement under treatment (i.e. stop of intravenous insulin treatment) up to a maximum of 14d

CONTACTS AND LOCATIONS:
Overall Officials: Marco Maggiorini, Prof. Dr. med., Principal Investigator — University Hospital Zürich, Department of Internal Medicine
Locations (1):
- University Hospital Zürich, Zurich, Switzerland